CLINICAL TRIAL: NCT06635213
Title: Determination of the Effectiveness of Desensitisation and Pain Neuroscience Training in Patients With Carpal Tunnel Syndrome With Nosiplastic Pain Phenotype
Brief Title: Effectiveness of Desensitisation and Pain Neuroscience Education in Patients With Carpal Tunnel Syndrome With Nosiplastic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Emrah Afsar, Phd, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024-b
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: After determining the predominant pain phenotype in patients with CTS, patients with mixed type (neuropathic and nosiplastic pain phenotype) will be randomly divided into two groups. One group (Group 1) will receive desensitisation and the other group (Group 2) will receive desensitisation and pain neuroscience education.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (desensitisation) (Active Comparator): Group 1 will receive desensitisation.
  Interventions: Other: Desensitisation
- Group 2 (desensitisation and pain neuroscience education) (Active Comparator): Group 2 will receive desensitisation and pain neuroscience education.
  Interventions: Other: Desensitisation; Other: Pain neuroscience education

INTERVENTIONS:
Other: Desensitisation — This technique is utilized to decrease, or normalize, the body's response to particular sensations.
Other: Pain neuroscience education — PNE is an educational intervention aiming to alter a patient's beliefs and cognitions regarding their pain experience.
  Arms: Group 2 (desensitisation and pain neuroscience education)

SUMMARY:
The aim of our study was to determine the effectiveness of desensitisation and pain neuroscience education in a group of patients with mixed phenotype pain (neuropathic and nosiplastic).

DETAILED DESCRIPTION:
People between the ages of 18-65, diagnosed with Carpal Tunnel Sedrome, who are suitable for the Nosiplastic pain phenotype and who volunteer to participate in the study will be included. The 7 steps in the Clinical Criteria/Rating System determined by the International Association for the Study of Pain (IASP) for Nosiplastic Pain will be applied to patients with CTS. After determining the predominant pain phenotype in patients with CTS, patients with mixed type (neuropathic and nosiplastic pain phenotype) will be randomly divided into two groups. One group (Group 1) will receive desensitisation and the other group (Group 2) will receive desensitisation and pain neuroscience education. Numerical rating scale (NRS) will be used for pain assessment. Boston Carpal Tunnel Questionnaire - Symptom Severity Scale will be used for symptom severity assessment and Boston Carpal Tunnel Questionnaire - Functional Status Scale will be used for functional status assessment. Pressure pain threshold will be measured with an algometer to evaluate hypersensitivity. The Pain Catastrophising Scale and the Tampa Kinesiophobia Scale will be administered to the patients. Normality of the data distribution will be assessed using the Shapiro-Wilk test. Fischer's exact test and chi-square test will be used to verify the relationship between categorical variables. A mixed model ANOVA will be performed on 2 (group 1 and group 2) x 3 (time: baseline, post-intervention, 3 months post-intervention) different outcome measures (pain intensity, symptom severity, functional status, pain catastrophising and kinesiophobia) to detect between-group differences.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with CTS
* Being suitable for the nosiplastic pain phenotype
* Being between the ages of 18-65
* Volunteering to participate in the study

Exclusion Criteria:

* Having systemic inflammatory disease
* Having a disease that may cause polyneuropathy such as diabetes mellitus
* Having a pacemaker
* Having a disease affecting the central nervous system
* Having cervical radiculopathy
* History of previous operation or local steroid injection due to CTS
* Hypersensitivity to heat and cold

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
Pressure Paın Threshold Measurement | [at the beginning of the study] [At the end of 6 weeks] [3 months later]
  The pressure pain threshold (PPT), the minimum amount of pressure at which the pressure sensation changes to pain, is measured with an electronic algometer (median nerve, ulnar nerve and radial nerve, C5-C6 zygapophyseal joint level (proximal), and tibialis anterior). Participants are asked to report when the sensation changes from pressure to pain. The mean of the three trials is calculated (with a 30 s rest interval in between).
Boston Carpal Tunnel Questionnaire - Symptom Severity Scale | [at the beginning of the study] [At the end of 6 weeks] [3 months later]
  Boston Carpal Tunnel Questionnaire - Symptom Severity Scale is an 11-item questionnaire used to assess symptom severity in individuals with CTS. Each item is scored from 1 to 5. Scores range from 1 (no symptoms) to 5 (worst symptoms). The patient's symptom severity score is the average score of 11 items.
Boston Carpal Tunnel Questionnaire - Functional Status Scale | [at the beginning of the study] [At the end of 6 weeks] [3 months later]
  Boston Carpal Tunnel Questionnaire - Functional Status Scale is an 8-item questionnaire used to assess the functional status of patients with CTS. Each item is scored from 1 to 5. Scores range from 1 (no functional deficit) to 5 (worst possible function). The patient's functional status score is the average of all 8 items.
Pain Catastrophising Scale | [at the beginning of the study] [At the end of 6 weeks] [3 months later]
  The Catastrophising Pain Scale (PCS) is used to measure catastrophising in response to pain through 13 statements with four possible options from 1 "never" to 4 "always". Higher scores indicate greater catastrophised pain.
Tampa Kinesiophobia Scale | [at the beginning of the study] [At the end of 6 weeks] [3 months later]
  It is a 17-question scale. The scale has a 4-point Likert scale (1= Strongly disagree, 4= Strongly agree). After reversing items 4, 8, 12 and 16, a total score is calculated. The person receives a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Numerical Rating Scale | [at the beginning of the study] [At the end of 6 weeks] [3 months later]
  Patients rate the current pain intensity from 0 ("no pain") to 10 ("worst possible pain").

SECONDARY OUTCOMES:
Cold Pain Threshold | 2 minutes
  For cold pain threshold, ice cubes (-5°C) placed in a plastic bag will be placed on the patients' skin for 10 seconds. Increased sensory perception will be considered as gain of function. The intensity of pain will also be recorded on an NRS scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Hot Pain Threshold | 2 minutes
  Thermal pain perception will be tested using a 3 cm2 sized metal piece equal to (lab-QST thermode size). The metal parts will be heated to 45˚C for hot pain threshold. The metal pieces will be applied to the skin for 3 seconds. It will be determined whether the stimulus is painful (yes/no), and if painful, the intensity of the pain on a numerical rating scale (NRS) (0: no pain, 10: imaginably worse pain).
Pressure Pain Threshold | 3 minutes
  A digital algometer will be used to measure Pressure Pain Threshold levels. Pressure will be applied at a rate of approximately 30 kPa/s with the algometer placed perpendicular to the point of application. Participants will be instructed to report when the sensation changes from pressure to pain. The intensity of pain will also be recorded on an NRS scale ranging from 0 (no pain at all) to 10 (worst pain imaginable).
Mechanical Pain Threshold | 3 minutes
  Mechanical pain threshold: to be assessed with a toothpick and a von Frey filament (256 mN). Increased sensory perception will be considered to reflect gain of function. The intensity of pain will also be recorded on an NRS scale ranging from 0 (no pain at all) to 10 (worst pain imaginable).
Dynamic Mechanical Allodynia | 3 minutes
  Patients will be touched on the affected area and the control area with a brush, an ear stick and a piece of cotton wool. The assessment tools will be applied 4 times by drawing a cross of 2 strokes (length 5 cm) at an angle of 90˚C in each direction. For each stimulus (brush/ear swab/cotton swab), they will indicate (1) whether the stimulus was perceived as painful (yes/no) and (2) the pain intensity on the NRS-11 (0 no pain, 10 imaginably worse pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)